CLINICAL TRIAL: NCT00106340
Title: Vildagliptin Compared to Glimepiride in Combination With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals Corporation
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A2308
Record Dates: First submitted 2005-03-22; First posted 2005-03-23 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: vildagliptin; Drug: Metformin; Drug: Glimepiride matching placebo
- Glimepiride (Active Comparator)
  Interventions: Drug: glimepiride; Drug: Metformin; Drug: Vildagliptin matching placebo

INTERVENTIONS:
Drug: vildagliptin
  Other Names: LAF237, Galvus
  Arms: Vildagliptin
Drug: glimepiride
  Arms: Glimepiride
Drug: Metformin
Drug: Vildagliptin matching placebo
  Arms: Glimepiride
Drug: Glimepiride matching placebo
  Arms: Vildagliptin

SUMMARY:
Many people with type 2 diabetes cannot maintain target blood glucose levels when taking a single oral drug. The purpose of this study is to assess the long term safety and effectiveness of vildagliptin, an unapproved drug, compared to that of glimepiride in lowering overall blood glucose levels when added to metformin in people with type 2 diabetes not at target blood glucose levels on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* On a stable dose of metformin as defined by the protocol
* Body mass index (BMI) in the range 22-45
* Blood glucose criteria must be met

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Evidence of significant diabetic complications
* Evidence of serious cardiovascular complications
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3118 (Actual)
Dates: Start 2005-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05-20 (Actual)

PRIMARY OUTCOMES:
Time to HbA1c >8% | 2 year

SECONDARY OUTCOMES:
Change from baseline in HbA1c at 5 years | 2 years (amended)
Adverse event profile after 5 years of treatment | 2 years (amended)
Coefficient of failure for HbA1c from week 24 to 5 years | 2 years (amended)
Change from baseline in fasting plasma glucose at 5 years | 2 years (amended)
Change from baseline in body weight at 5 years | 2 years (amended)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Nuremberg, Germany

REFERENCES:
- See also: Results for CLAF237A2308 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2649